CLINICAL TRIAL: NCT00058578
Title: Autologous T-Cell Depleted Peripheral Blood Stem Cell Transplantation for the Treatment of Selected Patients With Systemic Sclerosis
Brief Title: Stem Cell Transplant to Treat Patients With Systemic Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Dist Serv Prof, Center for Gene Therapy, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H7157; Systemic Sclerosis
Record Dates: First submitted 2003-04-08; First posted 2003-04-09 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Cyclophosphamide; Mesna; Granulocyte Colony-Stimulating Factor; Leukapheresis; Whole-Body Irradiation

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: Mesna
Drug: G-CSF
Procedure: Leukopheresis
Procedure: Total Body Irradiation

SUMMARY:
Systemic Sclerosis is a disease that may be caused by the immune system reacting against skin and certain organs. It is possible, that by changing the immune system we can modify the progression of this disease.

Stem cells are created in the bone marrow. They mature into different types of blood cells that are needed including red blood cells, white blood cells, and platelets. In this study, we will stimulate the bone marrow to make extra stem cells. Next we will collect the stem cells, select specific cells, and store them. We will then give high dose chemotherapy that will destroy the patients immune system. We will then give back the selected stem cells we collected. We believe that these selected stem cells may be able to "re-create" the immune system without the portion that causes Systemic Sclerosis.

The purpose of this study is to try to discover if stem cell transplantation can help patients with Systemic Sclerosis. We will also try to learn what the side effects are of this treatment in patients with Systemic Sclerosis. We hope that this treatment will help to relieve the symptoms patients are experiencing, although we do not know if it will.

DETAILED DESCRIPTION:
Before the transplant the research participant will receive daily G-CSF (Neupogen) for 5-6 days. This medication will help to stimulate the production of white blood cells (WBC) that will be used for the stem cell transplant. The G-CSF will be given as an injection into the arm.

If G-CSF does not stimulate the stem cells sufficiently, the patient will receive a single dose of drug called cyclophosphamide (chemotherapy) intravenously (into a vein). This drug will cause the blood cell counts to fall. A drug called MESNA will also be given to help protect the bladder from the Cyclophosphamide. After completing chemotherapy, patients will be started on G-CSF again until blood cell counts reach a certain level, at which time the patient will undergo leukopheresis. Leukopheresis is a procedure where blood is removed from one arm, pumped into a machine where the white blood cells are separated from most of the other cells and then returned through the same needle or through a needle in the other arm. This procedure usually takes 3 to 4 hours a day for up to 4 days in a row, depending on how many cells are collected each time.

After collection of the white blood cells, special agents (called monoclonal antibodies) will be used in the laboratory to select out certain types of white blood cells (CD34+ cells). The blood cells will be separated on a machine which picks out stem cells.

After leukopheresis, patients will receive drugs called cyclophosphamide and Mesna. They will also receive a drug called Atgam and radiation treatment to the entire body. This treatment will kill most of the blood forming cells in the bone marrow. We will then give the CD34+ cells that were collected during leukopheresis.

After the transplant patients will be followed closely, the same as any patient who receives a stem cell transplant. This follow-up will involve blood tests to see how the body is recovering after the chemotherapy and radiation, and a bone marrow aspiration once a year for 2 years.

ELIGIBILITY:
Eligibility Criteria:

* Patients aged < 60 years
* Patients must have either one major or 2 minor criteria for systemic sclerosis as per the criteria developed during the Scleroderma Criteria Cooperative Study.
* Rapidly progressive diffuse skin disease without other organ involvement (at least one of the following):

  * Scl-70 positive
  * Rodnam Skin score 16
  * With/without U3RNP antibodies; RNA polymerases 1-111 OR
* Internal Organ Involvement (at least one of the following):

  * Renal Proteinuria > 500mg/dl
  * Creatinine clearance > 50ml/min.
  * Blood pressure controlled to ≤ 160/110
  * Interstitial lung disease on high resolution CT
  * Hypoxemia (pO2 > 70 mmHg)
  * FVC > 50%
  * DLCO > 45%
  * Cardiac Disease
  * Myocarditis
  * Pericarditis
  * Coronary Artery Ejection Fraction > 30%
* Patients must meet the following hematological parameters:

  * Have an ANC > 500/mm3
  * Have a platelet count > 120 x lO9/l
  * Have a hemoglobin > 10g/dl

Exclusion Criteria:

* Patients > 60 years
* Patients with pulmonary, cardiac, hepatic, or renal impairment which would limit their ability to receive cytoreductive therapy and compromise their survival. This should include patients with any of the following:

  * Severe Lung Disease
  * Hypoxemia (pO2 £70 mmHg)
  * FVC of < 50%
  * DLCO of < 45%
  * Cardiac Disease
  * Ejection fraction < 30%
  * Uncontrolled arrhythmias
  * Cor. Pulmonale
  * Pulmonary hypertension (mPAP >/=60 mmHg)
  * Loss of digits or vascular access secondary to Raynaud's ischemia
  * History of oliguric renal failure or episode of renal crisiswith Glomerular filtration rate < 50ml/min Creatinine. Weight loss > 20% baseline since first involvement of gastrointestinal tract (midgut); or any patient requiring hyperalimentation prior to transplant because of gut dysfunction related to systemic sclerosis
  * SGOT/bilirubin > 2 x UPN on 2 repeated tests
  * Has active uncontrolled infection
  * Is sero-positive for HIV
  * Has demonstrated lack of compliance with prior medical care
  * Has active malignancy
  * Life expectancy is severely limited by illness other than scleroderma
  * Has evidence of myelodysplasia or prior extensive chemotherapy
  * Has uncontrolled hypertension
  * Positive pregnancy test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 1999-06; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Locations (1):
- The Methodist Hospital, Houston, Texas, United States